CLINICAL TRIAL: NCT03505346
Title: 68 Ga-NODAGA-E[c(RGDγK)]2: Positron Emission Tomography Tracer for Imaging of Angiogenesis in Ischemic Heart Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Simon Bentsen, Medical doctor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUDRA-CT: 2017-002712-14
Record Dates: First submitted 2018-03-05; First posted 2018-04-23 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Chronic Ischemic Heart Disease
Keywords: Positron Emission Tomography; nuclear medicine; prognosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutanous coronary intervention(PCI) (Experimental): 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 administered IV. two times. 14-21 days before intervention and 30-35 days after intervention
  Interventions: Drug: 68Ga-NODAGA-E[c(RGDyK)]2
- Coronary artery bypass-graft(CABG) (Experimental): 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 administered IV. two times. 14-21 days before intervention and 30-35 days after interventionintervention
  Interventions: Drug: 68Ga-NODAGA-E[c(RGDyK)]2

INTERVENTIONS:
Drug: 68Ga-NODAGA-E[c(RGDyK)]2 — 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 administered IV.
  Other Names: RGD-PET

SUMMARY:
The aim is to examine the expression of αvβ3 integrin using a novel selective radiotracer in patients with chronich ischemic heart disease and investigate if it is a suitable tool for predicting myocardial recovery and thus prognosis after intervention.

DETAILED DESCRIPTION:
Ischemic heart disease is worldwide the single most frequent cause of death. The number of patients surviving acute myocardial injury is increasing due to improved acute treatment. However, after the initial repair, the tissue undergoes a remodeling phase to compensate for the damaged area. This re-modeling phase can change the structure end geometry of the heart resulting in lower ejection fraction, leading to cardiac dysfunction, which eventually leads to heart failure. Ischemic heart disease is most commently caused by arteriosclerosis of the coronary artery.

If chronic ischemic heart disease is left untreated, it will lead to symptoms to the patient. These symptons occur when the myocardiel oxygen demand exceeds the oxygen provided, due to coronary occlusion.

If the heart suffers from ischemia, the tissue reacts strongly to the hypoxia. The body will as a compensatory mechanism create new vessel to provide the tissue with oxygen. This is known as the biological process of angiogenesis. This complex process involves different angiogenic and pro-fibrotic transcription factors that initiate the restoration of capillaries by sprouting from the existing endothelial cells in response to hypoxia.

Integrin αvβ3 is a transmembrane cell surface receptor that is markedly upregulated in states of angiogenesis. It facilitates migration and proliferation and thereby allowing cells to respond to extracellular environment. Integrin αvβ3 is thus a key player in the angiogenic process. The integrin αvβ3 has a binding site for an RGD peptide (Arg-Gly-Asp motif) and this can be targeted by PET tracers.

RGD-based PET tracers have been shown to accumulate at the site of myocardial necrosis in both human and animal studies. The uptake before interventions may correlate to recovery of cardiac function and thus serve as a prognostic marker after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years
* Patient with known chornic ischemic Heart disease admitted to Rigshospitalet to either PCI og CABG

Exclusion Criteria:

* No prior history of Heart surgery
* Not treated with anti-angiogenic medicine
* Subject with pacemaker, cochlear implant or insulin pump
* Pregnancy
* Lactation
* Severe claustrophobia
* Severe obesity (weight above 140kg)
* Conversion from PCI to CABG
* If a subject is in the fertile age, a pregnancy test will be use prior to injection to the PET_tracer
* If a subject is having a severe allergic reaction to the PET-tracer, the person will be excluded for the rest of the trial
* If the PET-tracer is administered subcutaneous, the person will be excluded for the rest of the trial¨
* Type I or II diabetes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate myocardial angiogenesis | 30-35 days
  Analysing change in uptake of 68Ga-NODAGA-E[c(RGDyK)]2 Positron Emission Tomography after intervention

SECONDARY OUTCOMES:
Correlation between 68Ga-NODAGA-E[c(RGDyK)]2 and myocardial perfusion | 30-35 days
  Correlation between uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and change in myocardial perfusion after intervention using Rubidium 82 Positron Emission Tomography
Correlation between 68Ga-NODAGA-E[c(RGDyK)]2 and functional recovery | 30-35 days
  Correlation between uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and functional recovery using Magnetic Resonance after intervention
Correlatino between 68Ga-NODAGA-E[c(RGDyK)]2 and viability | 30-35 days
  Correlation between uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and viability using Flour-Deoxy-Glucose Positron Emission Tomography after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Department of Physiology, Nuclear Medicine and PET, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No